CLINICAL TRIAL: NCT06741033
Title: Comparing the Effect of Toe-in Gait Modification Along With Conventional Physiotherapy in People With Medial Knee Osteoarthritis
Brief Title: Comparing the Effect of Toe-in Gait Modification Along With Conventional Physiotherapy in People With Medial KO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MSRSW/Batch-Fall22/758
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group I (Experimental)
  Interventions: Diagnostic Test: Conventional physiotherapy
- Interventional group II (Active Comparator)
  Interventions: Combination Product: Toe-in gait modification

INTERVENTIONS:
Diagnostic Test: Conventional physiotherapy — Conventional physiotherapy of medial knee osteoarthritis patients: Isometric exercises, strengthening exercises, stretching exercises and electrotherapy.
  Arms: Interventional group I
Combination Product: Toe-in gait modification — A specific alteration in walking pattern where the toes are directed inward during walking. This modification should be clearly defined, including the degree of inward rotation of the foot and how it is taught and monitored in participants. Toe-in gait modification basically includes decrease foot progression angle from baseline through internal foot rotation. Participants are instructed to increase the Toe-in angle of their study limb by 5 degree and walk at least 5-10 minutes (progressed to 15-20 min after 4 week) with this progression angle.
  Arms: Interventional group II

SUMMARY:
Medial knee osteoarthritis (OA) remains a prevalent and debilitating condition, despite conventional physiotherapy interventions aimed at reducing pain and improving function. This study investigates the additional benefits of toe-in gait modification when combined with conventional physiotherapy in individuals with medial knee OA. Rooted in biomechanical theories suggesting that altering gait patterns can reduce medial knee load, this research employs a randomized controlled trial methodology.

DETAILED DESCRIPTION:
Participants are divided into two groups: one receiving conventional physiotherapy alone, and the other receiving a combination of conventional physiotherapy and toe-in gait modification. Outcomes are assessed over a 8-week period, focusing on pain levels and physical function. The significance of this study lies in its potential to enhance current treatment protocols, offering a more effective, non-invasive intervention to alleviate symptoms and improve the quality of life for those suffering from medial knee OA. The findings could inform clinical practices and pave the way for personalized rehabilitation strategies that incorporate gait modifications, ultimately reducing the healthcare burden associated with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of MKOA having Grade 1-3 (radiographic evidence of MKOA)
* Knee pain on most days of previous month. (The most symptomatic side will consider the study limb for participants with bilaterally eligible knees)
* Age > 45
* Ability to walk unaided for at least 25 min
* Gender eligibility both male and female

Exclusion Criteria:

* Severe MKOA (Grade 4)
* Lateral OA
* Patella femoral OA
* Previous or planned hip or knee surgery
* Hip or ankle arthritis
* Rheumatoid arthritis
* Severe valgus and varus alignment requiring the use of an assistive device and the inability to walk independently
* Neurological dysfunction

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
NUMERIC PAIN RATING SCALE (NPRS) | 12 Months
  The NPRS is 11-point numeric scale ranges from '0' representing "no pain" to '10' representing "pain as bad as you can imagine
WOMAC scale | 12 Months
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales (Pain, Stiffness, and Physical Function) The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of orthopedic and rehabilitation IOR garden town, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No